CLINICAL TRIAL: NCT00868270
Title: Urinary Cytokine Levels as a Prognostic Marker for Kidney Scarring After Pyelonephritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Hassan Jassar, MD, Pediatrics Dept. Hillel Yaffe Medical Center
Other Study IDs: HY55-08
Record Dates: First submitted 2009-03-22; First posted 2009-03-24 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Kidney Scarring Post-Febrile UTI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Children with UTIs

SUMMARY:
The prevalence of kidney scarring after UTI is approximately 5-57%. UTIs are caused mainly by bacteria that cause local and systemic immunological reaction that are accompanied by cytokines. These cytokines are a main factor in the inflammatory process. They are produced by leukocytes, macrophages, fibroblasts, endothelial cells and epithelial cells in the kidney tissue. Interleukin 6 and 8 (IL-6 IL-8) were found in high levels in the urine of children and adults who suffer from UTIs. Other studies on animals have found a relationship between inflammatory reaction and scarring in the kidney. We hypothesize that we will find a similar relationship between the level of IL-6, IL-8 in the urine during acute pyelonephritis in children and the probability of kidney scarring.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-7
* First episode febrile UTI

Exclusion Criteria:

* Recurrent UTI

Max Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children with UTIs
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
High prevalence of kidney scarring in children with high levels of urine interleukins | six months

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel